CLINICAL TRIAL: NCT03256968
Title: An Open Label N of 1 Study to Evaluate the Study and Efficacy of Long-Term Treatment With Ivacaftor in Combination With Ataluren (PTC124) in Subjects With Nonsense Mutation Cystic Fibrosis
Brief Title: PTC Study to Evaluate Ataluren in Combination With Ivacaftor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Steven M Rowe, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F160106006
Record Dates: First submitted 2017-08-18; First posted 2017-08-22 (Actual); Results first posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ataluren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ataluren administration (Experimental): dose of the drug administered (mg/kg body weight)
  Interventions: Drug: Ataluren

INTERVENTIONS:
Drug: Ataluren — ataluren

SUMMARY:
The purpose of this study is to explore the combination of ataluren and ivacaftor as a treatment for patients with nonsense mutation cystic fibrosis

DETAILED DESCRIPTION:
Cystic Fibrosis (CF) is a life threatening genetic disorder resulting from mutations found in the CF gene known as the cystic fibrosis transmembrane conductance regulator or CFTR. This defect prevents correct chloride absorption in and out of the cells The purpose of this study is to explore the combination of ataluren and ivacaftor as a treatment for patients with a specific cystic fibrosis mutation

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of signed and dated informed consent/assent document(s) indicating that the subject (and/or his parent/legal guardian) has been informed of all pertinent aspects of the trial.
2. Age ≥6 years
3. Body weight ≥16 kg
4. Diagnosis of cystic fibrosis and documentation of the presence of a nonsense mutations of the CFTR gene, as determined by historical genotyping
5. Ability to perform a valid, reproducible spirometry with demonstration of a forced expiratory volume in 1second (FEV1) ≥30% and ≤90% of predicted for age, gender, and height.
6. If the subject is sexually active, willingness to abstain from sexual intercourse or employ a barrier or medical method of contraception during the study drug administration
7. Willingness and ability to comply with all study procedures and assessments.
8. Currently being administered ivacaftor, either alone (Kalydeco) or in combination with lumacaftor (Orkambi)

Exclusion Criteria:

1. Any change (initiation, change in type of drug, dose modification, schedule modification, interruption, discontinuation, or re-initiation) in a chronic treatment/prophylaxis regimen for CF or for CF-related conditions within 2 weeks prior to screening.
2. Ongoing participation in any other therapeutic clinical trial.
3. Evidence of pulmonary exacerbation or acute upper or lower respiratory tract infection (including viral illnesses) within 2 weeks prior to screening.
4. Ongoing inhaled tobramycin therapy.
5. Ongoing immunosuppressive therapy (other than corticosteroids up to 10mg/d equivalent of prednisone)
6. Ongoing warfarin, phenytoin, or tolbutamide therapy.
7. History of solid organ or hematological transplantation.
8. A history of positive hepatitis B surface antigen test, hepatitis C antibody test, or human immunodeficiency
9. Major complications of lung disease (including massive hemoptysis, pneumothorax, or pleural effusion) within 4 weeks prior to screening.
10. Pregnancy or breast-feeding.
11. Current smoker or a smoking history of ≥10 pack-years (number of cigarette packs/day × number of years smoked).
12. Prior or ongoing medical condition (eg, renal failure, alcoholism, drug abuse, psychiatric condition), medical history, physical findings, ECG findings, or laboratory abnormality that, in the investigator's opinion, could adversely affect the safety of the subject, makes it unlikely that the course of treatment or follow-up would be completed, or could impair the assessment of study results.

    -

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Rowe, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ataluren Administration
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ataluren Administration
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 31 [31 to 31]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: FEV1 as a Measure of Lung Function
Description: effect of ataluren on lung function as assessed by spirometry and measured by percentage of Liters (minimum value would be .0% Liters and maximum value of liters is dependent from person to person). The higher the value the better the outcome. The measure will include the change from baseline to one year to report a change between the two measurement points
Time Frame: 1 year
Measure: Number; unit: percentage of liters
Arm/Group | Ataluren Administration
Number analyzed (Participants) | 1
percentage of liters | .35

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Ataluren Administration
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ataluren Administration (N=1)
increased cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/68/NCT03256968/Prot_SAP_000.pdf